CLINICAL TRIAL: NCT04732962
Title: The Effect of a Biomechanical Footwear as a Non-invasive Alternative to Total Knee Replacement and as an Additional Rehabilitation Regimen Postoperatively
Brief Title: Biomechanical Footwear as a Non-invasive Alternative and Supplement to Total Knee Replacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Apos Medical and Sports Technology Ltd. (Industry)
Responsible Party: Principal Investigator, Michael Suk, MD, JD, MPH, MBA, FACS, Professor and Chair, Musculoskeletal Institute & Department of Orthopaedic Surgery, Geisinger Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0935
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- AposHealth (Experimental): Following the initial consultation and calibration of the Apos device in the clinic, the patients will receive from his therapist a home-based treatment plan. This usually includes wearing the device for about 20 minutes with about 20% of weight-bearing (patient is instructed to wear the Apos and just be with the device and go about his/her daily routine). A gradual increase in usage time is prescribed reaching up to 60 min wear time with about 40% weight-bearing.
  Patients are requested to return to follow-up (FU) appointments after 1, 3, 6, 9 and 12 months. In addition, patients will have a remote FU after 1-week to confirm they use AposHealth as advised. During the follow-up appointment, re-assessment of clinical outcomes and gait patterns are performed and the calibration of the Apos device is adjusted as needed. The treatment plan is adjusted, and patients are encouraged to continue to wear the device regularly at home.
  Interventions: Device: AposHealth
- Total Knee Replacement (TKR) (Active Comparator): Patients will undergo TKR according to Geisinger's policy, guidelines and care protocol.
  The study baseline visit will occur 6 weeks postoperative for TKR groups.
  Interventions: Procedure: Total Knee Replacement (TKR)
- Post TKR traditional physical therapy (PT) and AposHealth (Experimental): Patients who have had a knee replacement and were assigned to the traditional PT+ AposHealth group will follow Geisinger post-operative rehab protocol and will also receive AposHealth and follow the rehabilitation protocol.
  AposHealth will start six weeks post-op and will continue for 12 months. Patients will receive AposHealth similar to the non-invasive group, i.e., will have an initial evaluation (IE) and calibration of the Apos device, have a remote FU after one week from IE and in-clinic FUs at 1, 3 6, 9 and 12 months.
  Interventions: Device: AposHealth; Procedure: Total Knee Replacement (TKR)

INTERVENTIONS:
Device: AposHealth — AposHealth is comprised of a unique footwear (Apos device) and uses two convex pods called "Pertupods", which are screwed into the plantar surface of the sole so that a person walks on these pods. A trained Apos therapist calibrates the devices. The location of the pods is adjusted according to the treatment methodology, depending on the needed effect on unloading the knee and with the purpose of potentially alleviating pain immediately.
  Arms: AposHealth; Post TKR traditional physical therapy (PT) and AposHealth
Procedure: Total Knee Replacement (TKR) — A total knee replacement occurs when a diseased or damaged knee joint is totally replaced with an artificial joint called an implant. The implant consists of high-grade metal and plastic components that fuse to the resurfaced bone. It is designed to move like a healthy human joint.
  Arms: Post TKR traditional physical therapy (PT) and AposHealth; Total Knee Replacement (TKR)

SUMMARY:
Osteoarthritis (OA), the most common type of arthritis, affects more than 32.5 million adults in the United States. It is also among the most expensive condition to treat when joint replacement surgery is required. Although biomechanics plays an important role in OA disease, the non-surgical treatment options addressing biomechanics are scarce with limited effect. AposHealth is the fist biomechanical treatment that was shown to have a significant short-term effect on patients with knee OA.

The main objectives of this study are:

1. To assess AposHealth, a non-invasive home-based biomechanical treatment, as an alternative treatment for patients who are eligible for Total Knee Replacement (TKR).
2. To assess AposHealth as a new post-operative rehabilitation tool for patients post TKR.

DETAILED DESCRIPTION:
Osteoarthritis (OA), the most common type of arthritis, affects more than 32.5 million adults in the United States. It is also among the most expensive condition to treat when joint replacement surgery is required. Future projections of the prevalence of OA predict an increase in prevalence, mainly due to the aging of the population and obesity.

Total knee replacement (TKR) is the end-stage solution for patients with knee OA. The total annual cost of arthritis in the U.S. in 2013 reached over $300 billion. Expenditure is expected to grow significantly in response to the increase in prevalence and the projected number of TKRs.

Successful and beneficial non-invasive treatment options for knee OA are limited. More specifically, although biomechanics plays an important role in OA disease, the non-surgical treatment options addressing biomechanics are scarce with limited effect. AposHealth is the fist biomechanical treatment that was shown to have a significant short-term effect on patients with knee OA.

The main objectives of this study are:

1. To assess AposHealth, a non-invasive home-based biomechanical treatment, as an alternative treatment for patients who are eligible for TKR.
2. To assess AposHealth as a new post-operative rehabilitation tool for patients post TKR.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant women
* Between ages 45 and 80, inclusive
* ACR clinical criteria for OA of the knee
* Symptomatic uni- or bilateral OA of the knee for at least six months
* Radiological criteria: X-rays showing tibiofemoral knee osteoarthritis defined as at least Kellgren and Lawrence Grade 2
* At least a moderate NPRS pain score at baseline (≥5)
* Score of 1-3 based on the American Society of Anesthesiologists Physical Status Classification System
* Willing and able to read, comprehend, and sign the study informed consent form in English prior to study specific procedure

Exclusion Criteria:

* Body Mass Index (BMI) > 40
* History of an inflammatory rheumatic disease
* Non-knee musculoskeletal pain that is more severe than the knee pain
* Corticosteroids injections in the knees in the previous 6 weeks
* Previous major surgery to the knee such as osteotomy, hemiprosthesis, unilateral total joint replacement excluding knee arthroscopy > 6 months
* Patients with Geisinger Health Plan insurance for whom Apos is a covered treatment
* Patients with a recent history (<3 months) of a mental health condition, such as depression or anxiety
* Problems with balance (>2 unexplained falls within the last 12 months; experiencing regular dizziness that has caused a trip or fall; using a walking aid to get around such as a rollator, cane, walker)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
pain: Numerical Pain Rating Scale | 12 months
  score range: worst 0 - 10 best

SECONDARY OUTCOMES:
Veterans RAND 12 Health Survey (VR-12) physical component score | 3, 6, and 12 months
  patient's overall perspective of their physical health; worst 15 - 63 best
Koos Jr | 3, 6, and 12 months
  short form of knee injury and osteoarthritis outcome questionnaire; worst 0 - 100 best
pain: Numerical Pain Rating Scale | 3 and 6 months
  score range: worst 0 - 10 best
Step length (left and right) | 6 and 12 months
  A computerized mat is used to measure spatiotemporal gait parameters (ProtoKinetics Zeno™ Walkway Gait Analysis System). The gait mat detects pressure data during gait, during balance, and additional movement protocols. During the gait test, all patients are asked to walk barefoot at a self-selected speed. Patients walk 3 meters before and after the walkway mat to allow sufficient acceleration and deceleration time outside the measurement area. Each gait test included 6 walks and the mean value of the 6 walks is calculated for step length (in centimeters).
Single limb support (SLS): % gait cycle (left and right) | 6 and 12 months
  A computerized mat is used to measure spatiotemporal gait parameters (ProtoKinetics Zeno™ Walkway Gait Analysis System). The gait mat detects pressure data during gait, during balance, and additional movement protocols. During the gait test, all patients are asked to walk barefoot at a self-selected speed. Patients walk 3 meters before and after the walkway mat to allow sufficient acceleration and deceleration time outside the measurement area. Each gait test included 6 walks and the mean value of the 6 walks is calculated. A single gait cycle is defined from heel strike of one limb to the next heel strike (of the mane limb). A gait cycle is comprised of 2 phases: Stance (limb on the ground) and swing (limb swings forward). The stance phase is divided into SLS (one limb is on the ground while the other limb swings forward) and double limb support (both feet are on the ground). The absolute time of SLS will be converted to percent of gait cycle for standardization purposes.
Gait velocity | 6 and 12 months
  A computerized mat is used to measure spatiotemporal gait parameters (ProtoKinetics Zeno™ Walkway Gait Analysis System). The gait mat detects pressure data during gait, during balance, and additional movement protocols. During the gait test, all patients are asked to walk barefoot at a self-selected speed. Patients walk 3 meters before and after the walkway mat to allow sufficient acceleration and deceleration time outside the measurement area. Each gait test included 6 walks and the mean value of the 6 walks is calculated for velocity (meter/second).
Symmetry index (SI) for step length | 6 and 12 months
  A computerized mat is used to measure spatiotemporal gait parameters (ProtoKinetics Zeno™ Walkway Gait Analysis System). The gait mat detects pressure data during gait, during balance, and additional movement protocols. During the gait test, all patients are asked to walk barefoot at a self-selected speed. Patients walk 3 meters before and after the walkway mat to allow sufficient acceleration and deceleration time outside the measurement area. Each gait test included 6 walks and the mean value of the 6 walks is calculated for step length (in centimeters).
  Temporal distance (T-D) symmetry is used to calculate Symmetry Index (SI) for step length using the formula: (involved-uninvolved)/[(involved+uninvolved)/2)] x 100. SI value of zero represents perfect symmetry and up to 5% difference between limbs is considered normal.
Symmetry index (SI) for single limb support (SLS) | 6 and 12 months
  A computerized mat is used to measure spatiotemporal gait parameters (ProtoKinetics Zeno™ Walkway Gait Analysis System). Each gait test included 6 walks and the mean value is calculated. A single gait cycle is defined from heel strike of one limb to the next heel strike (of the mane limb). A gait cycle is comprised of 2 phases: Stance (limb on the ground) and swing (limb swings forward). The stance phase is divided into SLS (one limb is on the ground while the other limb swings forward) and double limb support (both feet are on the ground). The absolute time of SLS will be converted to % of gait cycle for standardization purposes. Temporal distance (T-D) symmetry is used to calculate Symmetry Index (SI) for SLS (% gait cycle) using the formula: (involved-uninvolved)/[(involved+uninvolved)/2)] x 100. SI value of zero represents perfect symmetry and up to 5% difference between limbs is considered normal.
Decay rate in AposTherapy group | 12 months
  Number of patients assigned to AposTherapy only group who schedule a TKR before end of study period
Pain medication intake | 3, 6, and 12 months
  Self-reported daily total milligrams of analgesic medication consumed

CONTACTS AND LOCATIONS:
Overall Officials: Michael Suk, MD, Principal Investigator — Geisinger Clinic
Locations (2):
- United States (2):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger - Orthopaedics Wilkes-Barre, Wilkes-Barre, Pennsylvania

IPD SHARING:
Plan to Share IPD: No